CLINICAL TRIAL: NCT05807945
Title: Comparison of the Effect of Intra-articular Administration of 0.2% Ropivacaine vs. 0.75% Ropivacaine as an Analgesic in the Immediate Postoperative Period of Knee Arthroscopy in Acute Injuries at the ABC Medical Center
Brief Title: "Comparison of Intra-articular of 0.2% Ropivacaine vs. 0.75% Ropivacaine in Postoperative of Knee Arthroscopy"
Acronym: ropivacaine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Paola M Zamora Munoz (Other)
Responsible Party: Sponsor-Investigator, Paola M Zamora Munoz, Principal Investigator, American British Cowdray Medical Center
Organization: American British Cowdray Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 001230620
Record Dates: First submitted 2023-03-05; First posted 2023-04-11 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Knee Arthroscopy; Acute Pain
Keywords: Knee Arthroscopy; Acute Pain; Ropivacaine
MeSH Terms: conditions — Acute Pain | interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: After confirming that the patients meet the selection criteria, they are invited to participate in the study. Upon accepting through signed informed consent, the physician in charge of randomization (physician 1) is informed and the surgery scheduled. The day of the surgery, the physician in charge of randomization reports the maneuver to be received from the anesthesiologist (physician 2) in charge, who prepares the dose of ropivacaine and gives it to a physician blinded to the maneuver (physician 3); this physician applies the ropivacaine intraarticular to the patient. The level of pain is evaluated two hours after the end of surgery by a physician blinded to the maneuver the patient has received (physician 4), while the patient is in his room, and the presence of acute-moderate-severe pain (4-10 points) is evaluated by a visual analog scale (vas) while the patient is requested to flex and extend the knee.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking was performed once the patient agreed to participate; the physician in charge of randomization informs the anesthesiologist of the maneuver that corresponds to the patient programmed for surgery, who prepares the dose for the patient and hands it to the physician who applies the maneuver (who is blinded to the maneuver). All patients receive 10 ml of solution with different doses of ropivacaine, the application vehicles being equal in physical appearance. The physician who evaluate the outcome does not participate in the randomization, surgery or application of the maneuver, and remains blinded to the dose the patient receives, as does the patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ropivacaine 0.75% Injectable Solution (Experimental): The patients receive 10 ml of intraarticular solution in the knee (at the anatomical point at the level of the upper pole of the ball joint, under the iliotibial band), with different content of ropivacaine 0.75%; the vehicle for application presents the same physical appearance for all patients and is applied by previously standardized treating physicians.
  Interventions: Drug: Ropivacaine 0.75% Injectable Solution
- Ropivacaine 0.2% Injectable Solution (Active Comparator): The patients receive 10 ml of intraarticular solution in the knee (at the anatomical point at the level of the upper pole of the ball joint, under the iliotibial band), with different content of ropivacaine 0.2%; the vehicle for application presents the same physical appearance for all patients and is applied by previously standardized treating physicians.
  Interventions: Drug: Ropivacaine 0.2% Injectable Solution

INTERVENTIONS:
Drug: Ropivacaine 0.75% Injectable Solution — The patients receive 10 ml of intraarticular solution in the knee (at the anatomical point at the level of the upper pole of the ball joint, under the iliotibial band), with different content of ropivacaine 0.75%; the vehicle for application presents the same physical appearance for all patients and is applied by previously standardized treating physicians.
  Arms: Ropivacaine 0.75% Injectable Solution
Drug: Ropivacaine 0.2% Injectable Solution — The patients receive 10 ml of intraarticular solution in the knee (at the anatomical point at the level of the upper pole of the ball joint, under the iliotibial band), with different content of ropivacaine 0.2%; the vehicle for application presents the same physical appearance for all patients and is applied by previously standardized treating physicians.
  Arms: Ropivacaine 0.2% Injectable Solution

SUMMARY:
All patients with acute lesions that attend the orthopedic and trauma center of the ABC medical center are invited to participate in the study. Those that meet the inclusion criteria and later sign an informed consent are randomized to receive 10 ml of a solution with ropivacaine at 0.75% and 0.2% intraarticular for the first 5 minutes after the end of surgery (closing of surgical wounds). Both the patient, the physician who applies it and the evaluator of outcomes remain blinded to the dose of ropivacaine the patient receives.

Two hours after the end of the surgery, while the patient is in his room, the presence of pain is evaluated by a visual analog scale (VAS), while the patient is asked to flex and extend his knee. The result is quantified continuously, to later categorize the pain in none to slight pain (0-3 points) and moderate-severe pain (4-10 points). All the information is recorded on established forms in the clinical file (general data), that includes the variables of interest for the study, and is reported by the physicians after standardization of all those in charge with collecting information to comply with the conceptual and operative operationalization of the variables described in the research protocol. In addition to the evaluation of pain, the administration of opioids to patients for necessary reasons (presence of pain) by the physicians in charge is recorded.

It is hoped that, in patients with knee arthroscopy for acute lesion, there is a difference in the frequency of moderate-severe pain of 30% in the post-operative (frequency of 37.5% in patients with ropivacaine at 0.2% and frequency of 0.75% in patients with ropivacaine at 0.75%).

DETAILED DESCRIPTION:
In previous studies the prevalence of moderate-severe intensity pain in patients post knee arthroscopy is 71.2%, and the prevalence of acute pain in post-operative is 37.5%, surpassing the prevalence when compared with other surgical procedures of various specialties.

The administration of opioids is part of common practice in managing pain. However, it represents a risk for patients due to adverse effects and the high risk of dependence. It is necessary to seek alternatives that reduce the consumption of opioids in patients post knee arthroscopy.

Characteristics of the patients reported in other studies, such as sex, body mass index, sedentarism, the cause, duration and use of tourniquet in surgery, in addition to the type of lesion of articular cartilage and the presence of neuropathies, may influence in the presence of pain severity.

ELIGIBILITY:
Inclusion Criteria:

* Mental health: healthy (not taking any medication)
* Articular cartilage lesion Grade I, II or III by Outerbridge
* Elective knee surgery
* Patients with any of the following diagnoses:
* Simple meniscal lesion
* Lesion of a single knee (unilateral)

Exclusion Criteria:

* Neuromotor diseases (alterations in step, strength or sensitivity)
* History of knee surgery (orthopedic)
* Instability that includes knee ligament lesions
* Addictions
* Mental diseases in medical treatment
* Hepatic diseases
* Allergy to any of the medications used in the study
* Epidural or peridural anesthesia
* Chronic pain in treatment
* Postoperative drain of knee arthroscopy
* Pregnant or lactating

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- American British Cowdray Medical Center, Mexico City, Cuajimalpa, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schulze E, Westphal AH, Veenhuis M, de Kok A. Purification and cellular localization of wild type and mutated dihydrolipoyltransacetylases from Azotobacter vinelandii and Escherichia coli expressed in E. coli. Biochim Biophys Acta. 1992 Mar 27;1120(1):87-96. doi: 10.1016/0167-4838(92)90428-g. PMID 1554745
- [Background] Brattwall M, Jacobson E, Forssblad M, Jakobsson J. Knee arthroscopy routines and practice. Knee Surg Sports Traumatol Arthrosc. 2010 Dec;18(12):1656-60. doi: 10.1007/s00167-010-1266-2. Epub 2010 Sep 21. PMID 20857086
- [Background] Kim S, Bosque J, Meehan JP, Jamali A, Marder R. Increase in outpatient knee arthroscopy in the United States: a comparison of National Surveys of Ambulatory Surgery, 1996 and 2006. J Bone Joint Surg Am. 2011 Jun 1;93(11):994-1000. doi: 10.2106/JBJS.I.01618. PMID 21531866
- [Background] Hoofwijk DMN, Fiddelers AAA, Emans PJ, Joosten EA, Gramke HF, Marcus MAE, Buhre WFFA. Prevalence and Predictive Factors of Chronic Postsurgical Pain and Global Surgical Recovery 1 Year After Outpatient Knee Arthroscopy: A Prospective Cohort Study. Medicine (Baltimore). 2015 Nov;94(45):e2017. doi: 10.1097/MD.0000000000002017. PMID 26559300
- [Background] Tepolt FA, Bido J, Burgess S, Micheli LJ, Kocher MS. Opioid Overprescription After Knee Arthroscopy and Related Surgery in Adolescents and Young Adults. Arthroscopy. 2018 Dec;34(12):3236-3243. doi: 10.1016/j.arthro.2018.07.021. Epub 2018 Nov 2. PMID 30396797
- [Background] Kanai A, Osawa S, Suzuki A, Ozawa A, Okamoto H, Hoka S. Regression of sensory and motor blockade, and analgesia during continuous epidural infusion of ropivacaine and fentanyl in comparison with other local anesthetics. Pain Med. 2007 Oct-Nov;8(7):546-53. doi: 10.1111/j.1526-4637.2006.00174.x. PMID 17883739
- [Background] Chew HF, Evans NA, Stanish WD. Patient-controlled bupivacaine infusion into the infrapatellar fat pad after anterior cruciate ligament reconstruction. Arthroscopy. 2003 May-Jun;19(5):500-5. doi: 10.1053/jars.2003.50110. PMID 12724679
- [Background] Okoroha KR, Keller RA, Marshall NE, Jung EK, Mehran N, Owashi E, Moutzouros V. Liposomal Bupivacaine Versus Femoral Nerve Block for Pain Control After Anterior Cruciate Ligament Reconstruction: A Prospective Randomized Trial. Arthroscopy. 2016 Sep;32(9):1838-45. doi: 10.1016/j.arthro.2016.05.033. Epub 2016 Jun 24. PMID 27349715
- [Background] Casati A, Santorsola R, Aldegheri G, Ravasi F, Fanelli G, Berti M, Fraschini G, Torri G. Intraoperative epidural anesthesia and postoperative analgesia with levobupivacaine for major orthopedic surgery: a double-blind, randomized comparison of racemic bupivacaine and ropivacaine. J Clin Anesth. 2003 Mar;15(2):126-31. doi: 10.1016/s0952-8180(02)00513-5. PMID 12719052
- [Background] Daniels SD, Garvey KD, Collins JE, Matzkin EG. Patient Satisfaction With Nonopioid Pain Management Following Arthroscopic Partial Meniscectomy and/or Chondroplasty. Arthroscopy. 2019 Jun;35(6):1641-1647. doi: 10.1016/j.arthro.2019.03.028. Epub 2019 May 6. PMID 31072715
- [Background] Ozdemir N, Kaya FN, Gurbet A, Yilmazlar A, Demirag B, Mandiraci BO. Comparison of intraarticular bupivacaine and levobupivacaine with morphine and epinephrine for knee arthroscopy. Eurasian J Med. 2013 Jun;45(2):77-82. doi: 10.5152/eajm.2013.18. PMID 25610257
- [Background] Kaeding CC, Hill JA, Katz J, Benson L. Bupivacaine use after knee arthroscopy: pharmacokinetics and pain control study. Arthroscopy. 1990;6(1):33-9. doi: 10.1016/0749-8063(90)90094-t. PMID 2310448
- [Background] Xu CP, Li X, Wang ZZ, Song JQ, Yu B. Efficacy and safety of single-dose local infiltration of analgesia in total knee arthroplasty: a meta-analysis of randomized controlled trials. Knee. 2014 Jun;21(3):636-46. doi: 10.1016/j.knee.2014.02.024. Epub 2014 Mar 13. PMID 24704172
- [Background] Jacobson E, Forssblad M, Rosenberg J, Westman L, Weidenhielm L. Can local anesthesia be recommended for routine use in elective knee arthroscopy? A comparison between local, spinal, and general anesthesia. Arthroscopy. 2000 Mar;16(2):183-90. doi: 10.1016/s0749-8063(00)90034-3. PMID 10705331
- [Background] Zou Z, An MM, Xie Q, Chen XY, Zhang H, Liu GJ, Shi XY. Single dose intra-articular morphine for pain control after knee arthroscopy. Cochrane Database Syst Rev. 2016 May 3;2016(5):CD008918. doi: 10.1002/14651858.CD008918.pub2. PMID 27140500
- [Background] Heller GZ, Manuguerra M, Chow R. How to analyze the Visual Analogue Scale: Myths, truths and clinical relevance. Scand J Pain. 2016 Oct;13:67-75. doi: 10.1016/j.sjpain.2016.06.012. Epub 2016 Jul 27. PMID 28850536
- [Background] Sun XL, Zhao ZH, Ma JX, Li FB, Li YJ, Meng XM, Ma XL. Continuous Local Infiltration Analgesia for Pain Control After Total Knee Arthroplasty: A Meta-analysis of Randomized Controlled Trials. Medicine (Baltimore). 2015 Nov;94(45):e2005. doi: 10.1097/MD.0000000000002005. PMID 26559294
- [Background] Merivirta R, Aarimaa V, Aantaa R, Koivisto M, Leino K, Liukas A, Kuusniemi K. Postoperative fentanyl patch versus subacromial bupivacaine infusion in arthroscopic shoulder surgery. Arthroscopy. 2013 Jul;29(7):1129-34. doi: 10.1016/j.arthro.2013.04.018. PMID 23809446
- [Background] Boden BP, Fassler S, Cooper S, Marchetto PA, Moyer RA. Analgesic effect of intraarticular morphine, bupivacaine, and morphine/bupivacaine after arthroscopic knee surgery. Arthroscopy. 1994 Feb;10(1):104-7. doi: 10.1016/s0749-8063(05)80301-9. PMID 8166893
- [Background] Zhou Y, Yang TB, Wei J, Zeng C, Li H, Yang T, Lei GH. Single-dose intra-articular ropivacaine after arthroscopic knee surgery decreases post-operative pain without increasing side effects: a systematic review and meta-analysis. Knee Surg Sports Traumatol Arthrosc. 2016 May;24(5):1651-9. doi: 10.1007/s00167-015-3656-y. Epub 2015 Jun 7. PMID 26049805
- [Background] Geutjens G, Hambidge JE. Analgesic effects of intraarticular bupivacaine after day-case arthroscopy. Arthroscopy. 1994 Jun;10(3):299-300. doi: 10.1016/s0749-8063(05)80116-1. PMID 8086025
- [Background] Panigrahi R, Roy R, Mahapatra AK, Prasad A, Priyadarshi A, Palo N. Intra-articular Adjuvant Analgesics following Knee Arthroscopy: Comparison between Single and Double Dose Dexmedetomidine and Ropivacaine A Multicenter Prospective Double-blind Trial. Orthop Surg. 2015 Aug;7(3):250-5. doi: 10.1111/os.12182. PMID 26311100
- [Background] Sorensen TS, Sorensen AI, Strange K. The effect of intra-articular instillation of bupivacaine on postarthroscopic morbidity: a placebo-controlled, double-blind trial. Arthroscopy. 1991;7(4):364-7. doi: 10.1016/0749-8063(91)90005-i. PMID 1755884
- [Background] El Baz MM, Farahat TEM. Efficacy of Adding Dexmedetomidine to Intra-articular Levobupivacaine on Postoperative Pain after Knee Arthroscopy. Anesth Essays Res. 2019 Apr-Jun;13(2):254-258. doi: 10.4103/aer.AER_23_19. PMID 31198240
- [Background] Ng HP, Nordstrom U, Axelsson K, Perniola AD, Gustav E, Ryttberg L, Gupta A. Efficacy of intra-articular bupivacaine, ropivacaine, or a combination of ropivacaine, morphine, and ketorolac on postoperative pain relief after ambulatory arthroscopic knee surgery: a randomized double-blind study. Reg Anesth Pain Med. 2006 Jan-Feb;31(1):26-33. doi: 10.1016/j.rapm.2005.09.009. PMID 16418021
- [Background] Rokhtabnak F, Ale Bouyeh MR, Seyed Siamdust A, Masoomshahi M, Aghajani M. Comparison of the effects of intra-articular sole ropivacaine and combined ketorolac and ropivacaine for pain control after knee arthroscopy surgery. Br J Pain. 2015 Aug;9(3):149-56. doi: 10.1177/2049463714553312. PMID 26516571
- [Background] Mitra S, Kaushal H, Gupta RK. Evaluation of analgesic efficacy of intra-articular bupivacaine, bupivacaine plus fentanyl, and bupivacaine plus tramadol after arthroscopic knee surgery. Arthroscopy. 2011 Dec;27(12):1637-43. doi: 10.1016/j.arthro.2011.08.295. Epub 2011 Nov 1. PMID 22047926
- [Background] Li C, Qu J. Efficacy of dexmedetomidine for pain management in knee arthroscopy: A systematic review and meta-analysis. Medicine (Baltimore). 2017 Oct;96(43):e7938. doi: 10.1097/MD.0000000000007938. PMID 29068980
- [Background] Khanna A, Saxena R, Dutta A, Ganguly N, Sood J. Comparison of ropivacaine with and without fentanyl vs bupivacaine with fentanyl for postoperative epidural analgesia in bilateral total knee replacement surgery. J Clin Anesth. 2017 Feb;37:7-13. doi: 10.1016/j.jclinane.2016.08.020. Epub 2016 Dec 22. PMID 28235533
- [Background] Lintner S, Shawen S, Lohnes J, Levy A, Garrett W. Local anesthesia in outpatient knee arthroscopy: a comparison of efficacy and cost. Arthroscopy. 1996 Aug;12(4):482-8. doi: 10.1016/s0749-8063(96)90044-4. PMID 8864008
- [Background] Iwasaki K, Sudo H, Kasahara Y, Yamada K, Ohnishi T, Tsujimoto T, Iwasaki N. Effects of Multiple Intra-articular Injections of 0.5% Bupivacaine on Normal and Osteoarthritic Joints in Rats. Arthroscopy. 2016 Oct;32(10):2026-2036. doi: 10.1016/j.arthro.2016.02.011. Epub 2016 Apr 29. PMID 27132778
- [Background] Milano G. Editorial Commentary: New Perspectives on the Intra-articular Use of Local Anesthetics: Five Weekly Injections of 0.5% Bupivacaine Does Not Alter Articular Cartilage. Arthroscopy. 2016 Oct;32(10):2037-2038. doi: 10.1016/j.arthro.2016.07.003. PMID 27697183
- [Background] Ravnihar K, Barlic A, Drobnic M. Effect of intra-articular local anesthesia on articular cartilage in the knee. Arthroscopy. 2014 May;30(5):607-12. doi: 10.1016/j.arthro.2014.02.002. PMID 24725314

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ropivacaine 0.75% Injectable Solution | Ropivacaine 0.2% Injectable Solution
Started | 36 | 34
Completed | 36 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ropivacaine 0.75% Injectable Solution | Ropivacaine 0.2% Injectable Solution | Total
Number analyzed (Participants) | 36 | 34 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 34 | 70
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (12) | 38 (11) | 39 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 26 | 51
  Male | 11 | 8 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Latin American | 36 | 34 | 70
Region of Enrollment [Number; unit: participants]
  Mexico | 36 | 34 | 70
Body Mass Index [Count of Participants; unit: Participants]
  <25 kg/m² | 18 | 17 | 35
  OVERWEIGHT (25 kg/m² or more) | 18 | 17 | 35
Time of articular cartilage lesion evolution [Count of Participants; unit: Participants]
  <14 days | 31 | 28 | 59
  >14 days | 5 | 6 | 11
Physical Activity [Count of Participants; unit: Participants]
  Sedentary | 29 | 22 | 51
  Active | 7 | 12 | 19
Etiology of surgery [Count of Participants; unit: Participants]
  Trauma | 26 | 29 | 55
  Degenerative | 10 | 5 | 15
Outerbridge Clasification [Count of Participants; unit: Participants]
  I (Softening or swelling of the cartilage, without visible fissures or fragmentation). | 16 | 7 | 23
  II (Fissures less than 50% of the cartilage thickness, 1 mm or less in depth) | 15 | 19 | 34
  III (Fissures extending more than 50% of the cartilage thickness but without full loss, 1-2 mm) | 5 | 8 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Acute Pain (Visual Analogue Scale)
Description: The result is quantified continuously in a scale from 0 (No pain) to 10 (Worst pain imaginable) points. Acute pain is labeled of a value ≥4 points.
Time Frame: 2 hours postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Ropivacaine 0.75% Injectable Solution | Ropivacaine 0.2% Injectable Solution
Number analyzed (Participants) | 36 | 34
Participants | 10 | 29

2. Secondary Outcome: Number of Participants With Opioid Administration
Description: The administration of opioids in the first two hours of postoperative for necessary reasons (pain ≥4 points) is recorded by the physician in charge.
Time Frame: 2 hours postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Ropivacaine 0.75% Injectable Solution | Ropivacaine 0.2% Injectable Solution
Number analyzed (Participants) | 36 | 34
Participants | 7 | 12

ADVERSE EVENTS:
Time Frame: 2 hours
Arm/Group | Ropivacaine 0.75% Injectable Solution | Ropivacaine 0.2% Injectable Solution
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/34
Other Adverse Events (participants affected / at risk) | 0/36 | 0/34

LIMITATIONS AND CAVEATS:
The main limitation of our study consists in the fact that the evaluation of pain is not an objective variable;, it was not possible for us to evaluate pain over a longer period of follow-up, due to the out-patient nature of the surgery.Our study did not evaluate the pre-operative intensity of pain, which is a weakness; however, patients were classified according to the severity of articular cartilage injury, variable that correlates with pain intensity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-26): https://cdn.clinicaltrials.gov/large-docs/45/NCT05807945/Prot_SAP_000.pdf